CLINICAL TRIAL: NCT01045733
Title: A Prospective Contralateral Comparison of Corneal Aberrations in Subjects Undergoing Aspheric Lens Implantation With Concomitant LRI and Aspheric Toric IOL Implantation
Brief Title: A Comparison of Corneal Aberrations in Subjects With Contralateral AcrySof IQ Toric Intraocular Lens (IOL) and AcrySof IQ IOL With Limbal Relaxing Incision (LRI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: M-09-045
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Cataract; Astigmatism
Keywords: Cataract; Toric; IOL; AcrySof; LRI; Astigmatism
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- IQ Toric IOL (Experimental): AcrySof IQ Toric intraocular lens (IOL) randomly assigned to one eye, with AcrySof IQ Aspheric IOL with Limbal Relaxing Incision (LRI) procedure in the fellow eye for contralateral implantation.
  Interventions: Device: AcrySof IQ Toric IOL
- IQ Aspheric IOL + LRI (Active Comparator): AcrySof IQ Aspheric intraocular lens (IOL) with Limbal Relaxing Incision (LRI) procedure randomly assigned to one eye, with AcrySof IQ Toric IOL in the fellow eye for contralateral implantation
  Interventions: Device: AcrySof IQ Aspheric IOL; Procedure: Limbal Relaxing Incision (LRI)

INTERVENTIONS:
Device: AcrySof IQ Toric IOL — AcrySof IQ Toric intraocular lens implanted in the capsular bag of the eye during cataract surgery. The IOL is intended for the lifetime of the patient.
  Other Names: AcrySof IQ Toric IOL Model SN6AT3; AcrySof IQ Toric IOL Model SN6AT4; AcrySof IQ Toric IOL Model SN6AT5
  Arms: IQ Toric IOL
Device: AcrySof IQ Aspheric IOL — AcrySof IQ aspheric intraocular lens implanted in the capsular bag of the eye during cataract surgery. The IOL is intended for the lifetime of the patient.
  Other Names: AcrySof IQ Aspheric IOL Model SN60WF
  Arms: IQ Aspheric IOL + LRI
Procedure: Limbal Relaxing Incision (LRI) — An incision was made at the corneal-limbal junction during cataract surgery for the purpose of relaxing corneal curvature, ie., correcting astigmatism.
  Arms: IQ Aspheric IOL + LRI

SUMMARY:
The purpose of this study was to evaluate and compare postoperative corneal aberrations and visual parameters in patients contralaterally implanted with an AcrySof IQ Toric intraocular lens (IOL) and AcrySof IQ Aspheric IOL with concomitant limbal relaxing incision.

ELIGIBILITY:
Inclusion Criteria:

Ocular criteria must be met in both eyes.

* Willing and able to understand and sign an informed consent;
* Willing and able to attend postoperative examinations per protocol schedule;
* Have cataracts that require extraction followed by implantation of a posterior chamber intraocular lens and used as an on-label procedure;
* Free of disease(s)/condition(s) listed in the "Caution" section of the AcrySof IQ and AcrySof IQ Toric package inserts;
* Have regular, bowtie shaped corneal astigmatism and qualify for an SN6AT3, SN6AT4 or SN6AT5 Intraocular Lens (IOL) in both eyes;
* Have the second surgery at least one week following the first eye implant but not later than one month after the first implant.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Previous corneal surgery;
* Planned multiple procedures during cataract/IOL implantation surgery;
* Ocular disease and/or condition that may compromise study results;
* Pregnant or planning pregnancy during course of study;
* Other protocol-defined exclusion criteria may apply.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-12; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Corneal Aberration | Month 6 postoperative

SECONDARY OUTCOMES:
Visual Acuity | Month 6 postoperative
Corneal Cylinder | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States